CLINICAL TRIAL: NCT03765450
Title: Pharmacokinetics of Infliximab and Tumor Necrosis Factor Concentrations in Serum, Stool, and Colonic Mucosa in Acute Severe Ulcerative Colitis
Brief Title: Pharmacokinetics of IFX and TNF Concentrations in Serum, Stool, and Colonic Mucosa in Acute Severe Ulcerative Colitis
Acronym: PROTOS
Status: Active, not recruiting | Type: Observational
Sponsor: Alimentiv Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: RP1713
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Ulcerative Colitis
Keywords: ASUC; Infliximab; Optimal Dose; Optimal Frequency; Theraputic Drug Monitoring
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, stool, tissue, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Study: Patients with Acute Severe Ulcerative Colitis who are either a) biologic-naïve or b) biologic-experienced without a known history of anti-infliximab antibodies requiring infliximab infusion therapy as a part of standard of care.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Patients will receive infliximab at the discretion of their physician as part of standard of care.

SUMMARY:
This is an open-label, prospective, observational study with the primary objective to characterize the pharmacokinetics of infliximab in patients with Acute Severe Ulcerative Colitis.

DETAILED DESCRIPTION:
In Acute Severe Ulcerative Colitis (ASUC), drug exposure may be affected by intestinal protein loss leading to hypoalbuminemia and rapid clearance of infliximab (IFX). Importantly, 2 studies have associated the loss of IFX in stool with poor outcomes. Multiple observational studies have identified that patients with faster IFX clearance have worse clinical outcomes and higher rates of antidrug antibody formation. To better understand optimal dosing of IFX in ASUC, the pharmacokinetics of IFX in association with outcomes must be better defined in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Present to hospital with ASUC based on Truelove and Witts criteria,33 defined as the presence of more than 6 bloody stools per day along with any 1 of the following: tachycardia > 90 beats per minute, fever > 37.8 °C, hemoglobin < 10.5 g/dL, and erythrocyte sedimentation rate (ESR) > 30 mm/h (or CRP > 30 mg/L [high-sensitivity CRP > 300 mg/L]) is a suitable surrogate if ESR is not available1).
* Have a partial MCS > 7.
* Have a Mayo Clinic ES ≥ 2 with disease extending 15 cm or more beyond the anal verge.
* Require rescue inpatient IFX infusion as part of routine care. Note, the IFX treatment regimen is not defined by this protocol and any dosage regimen is acceptable for the purposes of this study, such as standard or accelerated induction regimens.
* Be able to speak English and participate fully in all aspects of this clinical trial.
* Provide written informed consent.

Exclusion Criteria:

* A known history of being positive for anti-IFX antibodies.
* Have a serious active infection, active malignancy, or any other known condition contraindicated with infliximab therapy, according to current prescribing information.
* Serious underlying disease other than ASUC, or other physical or psychosocial condition that, in the opinion of the investigator, may interfere with the subject's ability to participate fully in the study.
* Prior enrollment in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute severe ulcerative colitis, who are biologic-naive or biologic-experienced without a known history of anti-infliximab antibodies and will be receiving infliximab infusion therapy.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Inter-compartmental Difference in Infliximab Concentration | 22 weeks
  Infliximab population pharmacokinetics

SECONDARY OUTCOMES:
Change in Proteome | 22 weeks
  Change in Proteomics before and after therapy
Change in Transcriptome | 22 weeks
  Change in Transcriptomics before and after therapy
Change in Robarts Histopathologic Index | 22 weeks
  Change in Robarts Histopathologic Index before and after therapy The RHI consists of 4 histological items (extent of chronic inflammatory cell infiltration, neutrophils in the lamina propria, neutrophils in the epithelium, and erosions and ulceration) scored from 0 to 3 and multiplied by a weighting factor. The total RHI score is calculated by summing the weighted scores of the histological items, with total scores ranging from 0 (no disease activity) to 33 (severe disease activity).
Change in Mayo Clinic Endoscopic Score | 22 weeks
  Change in Mayo Clinic Endoscopic Score before and after therapy The Mayo Clinic score (MCS) scores 4 variables (stool frequency, rectal bleeding, a physician's global assessment and endoscopic findings with flexible sigmoidoscopy). The endoscopic component of the MCS assesses disease activity on a 4-point scale (0-3 points), with higher scores representing more severe disease activity. Mucosal healing is often defined as an endoscopy score of 0 or 1.
  Normal or inactive disease = 0 Mild disease (erythema, decreased vascular pattern, mild friability) = 1 Moderate disease (marked erythema, absent vascular pattern, friability, erosions) = 2 Severe (spontaneous bleeding, ulceration) = 3

CONTACTS AND LOCATIONS:
Overall Officials: Niels Vande Casteele, Study Director — UCSD
Locations (3):
- United States (2):
  - UCSD, San Diego, California
  - Cornell University, New York, New York
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Dinesen LC, Walsh AJ, Protic MN, Heap G, Cummings F, Warren BF, George B, Mortensen NJ, Travis SP. The pattern and outcome of acute severe colitis. J Crohns Colitis. 2010 Oct;4(4):431-7. doi: 10.1016/j.crohns.2010.02.001. Epub 2010 Feb 19. PMID 21122540
- [Background] Williams JG, Alam MF, Alrubaiy L, Clement C, Cohen D, Grey M, Hilton M, Hutchings HA, Longo M, Morgan JM, Rapport FL, Seagrove AC, Watkins A. Comparison Of iNfliximab and ciclosporin in STeroid Resistant Ulcerative Colitis: pragmatic randomised Trial and economic evaluation (CONSTRUCT). Health Technol Assess. 2016 Jun;20(44):1-320. doi: 10.3310/hta20440. PMID 27329657
- [Background] Seah D, De Cruz P. Review article: the practical management of acute severe ulcerative colitis. Aliment Pharmacol Ther. 2016 Feb;43(4):482-513. doi: 10.1111/apt.13491. Epub 2016 Jan 4. PMID 26725569
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Background] Sandborn WJ, Rutgeerts P, Feagan BG, Reinisch W, Olson A, Johanns J, Lu J, Horgan K, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Colectomy rate comparison after treatment of ulcerative colitis with placebo or infliximab. Gastroenterology. 2009 Oct;137(4):1250-60; quiz 1520. doi: 10.1053/j.gastro.2009.06.061. Epub 2009 Jul 28. PMID 19596014
- [Background] Jarnerot G, Hertervig E, Friis-Liby I, Blomquist L, Karlen P, Granno C, Vilien M, Strom M, Danielsson A, Verbaan H, Hellstrom PM, Magnuson A, Curman B. Infliximab as rescue therapy in severe to moderately severe ulcerative colitis: a randomized, placebo-controlled study. Gastroenterology. 2005 Jun;128(7):1805-11. doi: 10.1053/j.gastro.2005.03.003. PMID 15940615
- [Background] Sands BE, Tremaine WJ, Sandborn WJ, Rutgeerts PJ, Hanauer SB, Mayer L, Targan SR, Podolsky DK. Infliximab in the treatment of severe, steroid-refractory ulcerative colitis: a pilot study. Inflamm Bowel Dis. 2001 May;7(2):83-8. doi: 10.1097/00054725-200105000-00001. PMID 11383595
- [Background] Narula N, Marshall JK, Colombel JF, Leontiadis GI, Williams JG, Muqtadir Z, Reinisch W. Systematic Review and Meta-Analysis: Infliximab or Cyclosporine as Rescue Therapy in Patients With Severe Ulcerative Colitis Refractory to Steroids. Am J Gastroenterol. 2016 Apr;111(4):477-91. doi: 10.1038/ajg.2016.7. Epub 2016 Feb 9. PMID 26856754
- [Background] Gibson DJ, Heetun ZS, Redmond CE, Nanda KS, Keegan D, Byrne K, Mulcahy HE, Cullen G, Doherty GA. An accelerated infliximab induction regimen reduces the need for early colectomy in patients with acute severe ulcerative colitis. Clin Gastroenterol Hepatol. 2015 Feb;13(2):330-335.e1. doi: 10.1016/j.cgh.2014.07.041. Epub 2014 Jul 30. PMID 25086187
- [Background] Govani SM, Waljee AK, Stidham RW, et al. Accelerated dosing of infliximab prevents colectomy within 90 days in only half of patients with severe ulcerative colitis [abstract]. Gastroenterology. 2016;150:S106. Abstract no. 516.
- [Background] Al Khoury A, Chao C-y, Bessissow T, et al. Intensified infliximab rescue therapy for acute severe ulcerative colitis does not improve long term colectomy-free survival [abstract]. Gastroenterology. 2017;152:S399. Abstract no. P495.
- [Background] Choy MC, Seah D, Gorelik A, et al. Comparison of accelerated infliximab induction vs standard induction treatment in acute severe ulcerative colitis [abstract]. Gastroenterology. 2016;150:S803. Abstract no. Mo1878.
- [Background] Afif W, Loftus EV Jr, Faubion WA, Kane SV, Bruining DH, Hanson KA, Sandborn WJ. Clinical utility of measuring infliximab and human anti-chimeric antibody concentrations in patients with inflammatory bowel disease. Am J Gastroenterol. 2010 May;105(5):1133-9. doi: 10.1038/ajg.2010.9. Epub 2010 Feb 9. PMID 20145610
- [Background] Seow CH, Newman A, Irwin SP, Steinhart AH, Silverberg MS, Greenberg GR. Trough serum infliximab: a predictive factor of clinical outcome for infliximab treatment in acute ulcerative colitis. Gut. 2010 Jan;59(1):49-54. doi: 10.1136/gut.2009.183095. PMID 19651627
- [Background] Kevans D, Murthy S, Iacono A, et al. Accelerated clearance of serum infliximab during induction therapy for acute ulcerative colitis is associated with treatment failure [abstract]. Gastroenterology. 2012;142:S-384-S-385. Abstract no. Sa2031
- [Background] Papamichael K, Rivals-Lerebours O, Billiet T, Vande Casteele N, Gils A, Ferrante M, Van Assche G, Rutgeerts PJ, Mantzaris GJ, Peyrin-Biroulet L, Vermeire S. Long-Term Outcome of Patients with Ulcerative Colitis and Primary Non-response to Infliximab. J Crohns Colitis. 2016 Sep;10(9):1015-23. doi: 10.1093/ecco-jcc/jjw067. Epub 2016 Mar 28. PMID 27022161
- [Background] Arias MT, Vande Casteele N, Vermeire S, de Buck van Overstraeten A, Billiet T, Baert F, Wolthuis A, Van Assche G, Noman M, Hoffman I, D'Hoore A, Gils A, Rutgeerts P, Ferrante M. A panel to predict long-term outcome of infliximab therapy for patients with ulcerative colitis. Clin Gastroenterol Hepatol. 2015 Mar;13(3):531-8. doi: 10.1016/j.cgh.2014.07.055. Epub 2014 Aug 10. PMID 25117777
- [Background] Adedokun OJ, Sandborn WJ, Feagan BG, Rutgeerts P, Xu Z, Marano CW, Johanns J, Zhou H, Davis HM, Cornillie F, Reinisch W. Association between serum concentration of infliximab and efficacy in adult patients with ulcerative colitis. Gastroenterology. 2014 Dec;147(6):1296-1307.e5. doi: 10.1053/j.gastro.2014.08.035. Epub 2014 Aug 28. PMID 25173754
- [Background] Brandse JF, Mathot RA, van der Kleij D, Rispens T, Ashruf Y, Jansen JM, Rietdijk S, Lowenberg M, Ponsioen CY, Singh S, van den Brink GR, D'Haens GR. Pharmacokinetic Features and Presence of Antidrug Antibodies Associate With Response to Infliximab Induction Therapy in Patients With Moderate to Severe Ulcerative Colitis. Clin Gastroenterol Hepatol. 2016 Feb;14(2):251-8.e1-2. doi: 10.1016/j.cgh.2015.10.029. Epub 2015 Nov 9. PMID 26545802
- [Background] Papamichael K, Van Stappen T, Vande Casteele N, Gils A, Billiet T, Tops S, Claes K, Van Assche G, Rutgeerts P, Vermeire S, Ferrante M. Infliximab Concentration Thresholds During Induction Therapy Are Associated With Short-term Mucosal Healing in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2016 Apr;14(4):543-9. doi: 10.1016/j.cgh.2015.11.014. Epub 2015 Dec 8. PMID 26681486
- [Background] Brandse JF, van den Brink GR, Wildenberg ME, van der Kleij D, Rispens T, Jansen JM, Mathot RA, Ponsioen CY, Lowenberg M, D'Haens GR. Loss of Infliximab Into Feces Is Associated With Lack of Response to Therapy in Patients With Severe Ulcerative Colitis. Gastroenterology. 2015 Aug;149(2):350-5.e2. doi: 10.1053/j.gastro.2015.04.016. Epub 2015 Apr 25. PMID 25917786
- [Background] Brandse JF, Wildenberg M, De Bruyn JR, et al. Fecal loss of infliximab as a cause of lack of response in severe inflammatory bowel disease [abstract]. Gastroenterology. 2013;1:S36. Abstract no. 157.
- [Background] Frieri G, Giacomelli R, Pimpo M, Palumbo G, Passacantando A, Pantaleoni G, Caprilli R. Mucosal 5-aminosalicylic acid concentration inversely correlates with severity of colonic inflammation in patients with ulcerative colitis. Gut. 2000 Sep;47(3):410-4. doi: 10.1136/gut.47.3.410. PMID 10940280
- [Background] Yarur AJ, Jain A, Sussman DA, Barkin JS, Quintero MA, Princen F, Kirkland R, Deshpande AR, Singh S, Abreu MT. The association of tissue anti-TNF drug levels with serological and endoscopic disease activity in inflammatory bowel disease: the ATLAS study. Gut. 2016 Feb;65(2):249-55. doi: 10.1136/gutjnl-2014-308099. Epub 2015 Feb 10. PMID 25670812
- [Background] Olsen T, Cui G, Goll R, Husebekk A, Florholmen J. Infliximab therapy decreases the levels of TNF-alpha and IFN-gamma mRNA in colonic mucosa of ulcerative colitis. Scand J Gastroenterol. 2009;44(6):727-35. doi: 10.1080/00365520902803507. PMID 19294580
- [Background] Hartman DS, Tracey DE, Lemos BR, Erlich EC, Burton RE, Keane DM, Patel R, Kim S, Bhol KC, Harris MS, Fox BS. Effects of AVX-470, an Oral, Locally Acting Anti-Tumour Necrosis Factor Antibody, on Tissue Biomarkers in Patients with Active Ulcerative Colitis. J Crohns Colitis. 2016 Jun;10(6):641-9. doi: 10.1093/ecco-jcc/jjw026. Epub 2016 Jan 22. PMID 26802087
- [Background] Toedter G, Li K, Marano C, Ma K, Sague S, Huang CC, Song XY, Rutgeerts P, Baribaud F. Gene expression profiling and response signatures associated with differential responses to infliximab treatment in ulcerative colitis. Am J Gastroenterol. 2011 Jul;106(7):1272-80. doi: 10.1038/ajg.2011.83. Epub 2011 Mar 29. PMID 21448149
- [Background] West NR, Hegazy AN, Owens BMJ, Bullers SJ, Linggi B, Buonocore S, Coccia M, Gortz D, This S, Stockenhuber K, Pott J, Friedrich M, Ryzhakov G, Baribaud F, Brodmerkel C, Cieluch C, Rahman N, Muller-Newen G, Owens RJ, Kuhl AA, Maloy KJ, Plevy SE; Oxford IBD Cohort Investigators; Keshav S, Travis SPL, Powrie F. Oncostatin M drives intestinal inflammation and predicts response to tumor necrosis factor-neutralizing therapy in patients with inflammatory bowel disease. Nat Med. 2017 May;23(5):579-589. doi: 10.1038/nm.4307. Epub 2017 Apr 3. PMID 28368383
- [Background] Sands BE, Chen J, Feagan BG, Penney M, Rees WA, Danese S, Higgins PDR, Newbold P, Faggioni R, Patra K, Li J, Klekotka P, Morehouse C, Pulkstenis E, Drappa J, van der Merwe R, Gasser RA Jr. Efficacy and Safety of MEDI2070, an Antibody Against Interleukin 23, in Patients With Moderate to Severe Crohn's Disease: A Phase 2a Study. Gastroenterology. 2017 Jul;153(1):77-86.e6. doi: 10.1053/j.gastro.2017.03.049. Epub 2017 Apr 5. PMID 28390867
- [Background] Bloemendaal FM, Levin AD, Wildenberg ME, Koelink PJ, McRae BL, Salfeld J, Lum J, van der Neut Kolfschoten M, Claassens JW, Visser R, Bentlage A, D'Haens GRAM, Verbeek JS, Vidarsson G, van den Brink GR. Anti-Tumor Necrosis Factor With a Glyco-Engineered Fc-Region Has Increased Efficacy in Mice With Colitis. Gastroenterology. 2017 Nov;153(5):1351-1362.e4. doi: 10.1053/j.gastro.2017.07.021. Epub 2017 Jul 27. PMID 28756234
- [Background] Bhol KC, Tracey DE, Lemos BR, Lyng GD, Erlich EC, Keane DM, Quesenberry MS, Holdorf AD, Schlehuber LD, Clark SA, Fox BS. AVX-470: a novel oral anti-TNF antibody with therapeutic potential in inflammatory bowel disease. Inflamm Bowel Dis. 2013 Oct;19(11):2273-81. doi: 10.1097/MIB.0b013e3182a11958. PMID 23949620
- [Background] Harris MS, Hartman D, Lemos BR, Erlich EC, Spence S, Kennedy S, Ptak T, Pruitt R, Vermeire S, Fox BS. AVX-470, an Orally Delivered Anti-Tumour Necrosis Factor Antibody for Treatment of Active Ulcerative Colitis: Results of a First-in-Human Trial. J Crohns Colitis. 2016 Jun;10(6):631-40. doi: 10.1093/ecco-jcc/jjw036. Epub 2016 Jan 28. PMID 26822613
- [Background] TRUELOVE SC, WITTS LJ. Cortisone in ulcerative colitis; final report on a therapeutic trial. Br Med J. 1955 Oct 29;2(4947):1041-8. doi: 10.1136/bmj.2.4947.1041. No abstract available. PMID 13260656
- [Background] Schroeder KW, Tremaine WJ, Ilstrup DM. Coated oral 5-aminosalicylic acid therapy for mildly to moderately active ulcerative colitis. A randomized study. N Engl J Med. 1987 Dec 24;317(26):1625-9. doi: 10.1056/NEJM198712243172603. PMID 3317057
- [Background] Kennedy JJ, Whiteaker JR, Schoenherr RM, Yan P, Allison K, Shipley M, Lerch M, Hoofnagle AN, Baird GS, Paulovich AG. Optimized Protocol for Quantitative Multiple Reaction Monitoring-Based Proteomic Analysis of Formalin-Fixed, Paraffin-Embedded Tissues. J Proteome Res. 2016 Aug 5;15(8):2717-28. doi: 10.1021/acs.jproteome.6b00245. Epub 2016 Jul 27. PMID 27462933
- [Background] Willrich MA, Murray DL, Barnidge DR, Ladwig PM, Snyder MR. Quantitation of infliximab using clonotypic peptides and selective reaction monitoring by LC-MS/MS. Int Immunopharmacol. 2015 Sep;28(1):513-20. doi: 10.1016/j.intimp.2015.07.007. Epub 2015 Jul 25. PMID 26210595
- [Background] Vande Casteele N, Mould DR, Coarse J, Hasan I, Gils A, Feagan B, Sandborn WJ. Accounting for Pharmacokinetic Variability of Certolizumab Pegol in Patients with Crohn's Disease. Clin Pharmacokinet. 2017 Dec;56(12):1513-1523. doi: 10.1007/s40262-017-0535-3. PMID 28353055
- [Background] YOUDEN WJ. Index for rating diagnostic tests. Cancer. 1950 Jan;3(1):32-5. doi: 10.1002/1097-0142(1950)3:13.0.co;2-3. No abstract available. PMID 15405679